CLINICAL TRIAL: NCT02434107
Title: Controlled and Prospective Randomised Study to Compare Complete Lymph Node Dissection Versus Watchful Waiting in Patients With Malignant Melanoma With a Tumour Thickness of 1,0mm+ and Evidence of Metastases in the Sentinel Node
Brief Title: Complete Lymph Node Dissection vs Watchful Waiting in Patients With Malignant Melanoma (Thickness of 1,0mm+ and Evidence of Metastases in the Sentinel Node)
Acronym: DeCOG-SLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V1410112004
Record Dates: First submitted 2015-04-02; First posted 2015-05-05 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2017-05

CONDITIONS: Melanoma
Keywords: Sentinel Lymph Node Biopsy; Lymph Node Excision
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Completion Lymphadenectomy (Experimental): Completion Lymphadenectomy and monitoring afterwards
  Interventions: Procedure: Completion Lymphadenectomy
- Clinical Monitoring (Palpation and node ultrasound) (Experimental): Monitoring only
  Interventions: Procedure: Clinical Monitoring (Palpation and node ultrasound)

INTERVENTIONS:
Procedure: Completion Lymphadenectomy
  Arms: Completion Lymphadenectomy
Procedure: Clinical Monitoring (Palpation and node ultrasound)
  Arms: Clinical Monitoring (Palpation and node ultrasound)

SUMMARY:
Sentinel lymph node biopsy (SLNB) is considered as standard diagnostic procedure in melanoma patients carrying a reasonable risk for metastases. In numerous studies the prognostic role of micro metastases in the sentinel node (SN) was described. However, the prognostic value of a complete lymph node dissection in patients with a positive SN is still unclear.

This study was planned to analyse the survival outcome of patients with a positive SN receiving complete lymphadenectomy versus watchful waiting.

ELIGIBILITY:
Inclusion Criteria:

* Cutaneous melanoma with a tumour thickness of at least 1,00mm
* Positive sentinel node with micro metastases of max. 2mm in diameter

Exclusion Criteria:

* Mucosal or ocular melanoma
* Cutaneous melanoma located in the head/neck region
* Evidence of satellite, in transit or local metastases / recurrences
* Macro metastases of the SN or micro metastases of >2mm in diameter
* Additional immune-suppressive therapy
* Pregnant of lactating women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 483 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Distant metastases free survival | 3 Years

SECONDARY OUTCOMES:
Distant metastases free survival | 5 Years

CONTACTS AND LOCATIONS:
Overall Officials: Claus Garbe, MD, Study Director — University Hopsital Tübingen; Rudolf Stadler, MD, Study Chair — Johannes Wesling Klinikum Minden
Locations (41):
- Germany (41):
  - Humboldt-Universität Berlin Charité, Berlin
  - Krankenhaus Neukölln, Berlin
  - Universtitäts-Hautklinik Bochum, Bochum
  - Zentralkrankenhaus, Bremen
  - Universität Köln, Cologne
  - Carl-Thiem Klinikum, Cottbus
  - Städtische Kliniken Darmstadt, Darmstadt
  - Städtische Kliniken Dessau, Dessau
  - Städtisches Klinikum Friedrichsstadt, Dresden
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Heinrich Heine Universität, Düsseldorf
  - Klinikum Erfurt GmbH, Erfurt
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Klinkum der J. W. Goethe Universität, Frankfurt am Main
  - Klinikum der Albert-Ludwigs-Universität, Freiburg im Breisgau
  - Justus-Liebig-Universität, Giessen
  - Georg-August Universität, Göttingen
  - Allgemeines Krankenhaus St. Georg, Hamburg
  - Klinikum de Ruprecht-Karls-Universität, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Klinikum der Friedrich Schiller Universität, Jena
  - Städtische Hautklinik Karlsruhe, Karlsruhe
  - Städtische Kliniken Kassel, Kassel
  - Universität Leipzig, Leipzig
  - Klinkum Lippe-Lemgo GmbH, Lemgo
  - Universitätsklinikum Lübeck, Lübeck
  - Otto-von-Guericke-Universität, Magdeburg
  - Klinik der Philipps-Universität, Marburg
  - Johannes Wesling Klinikum Minden, Minden
  - Ludwig-Maximilians-Universität, Munich
  - Technische Universität, Munich
  - Städt. Krankenhaus München-Schwabing, Munich
  - Universitätsklinkum Münster, Münster
  - Städtische Kliniken Oldenburg, Oldenburg
  - Klinkum der Universität, Regensburg
  - Eberhard-Karls Universität, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Katholisches Krankenhaus, Unna
  - Klinkum Wuppertal GmbH, Wuppertal
  - Universitätsklinik und Poliklinik, Würzburg

REFERENCES:
- [Derived] Leiter U, Stadler R, Mauch C, Hohenberger W, Brockmeyer NH, Berking C, Sunderkotter C, Kaatz M, Schatton K, Lehmann P, Vogt T, Ulrich J, Herbst R, Gehring W, Simon JC, Keim U, Verver D, Martus P, Garbe C; German Dermatologic Cooperative Oncology Group. Final Analysis of DeCOG-SLT Trial: No Survival Benefit for Complete Lymph Node Dissection in Patients With Melanoma With Positive Sentinel Node. J Clin Oncol. 2019 Nov 10;37(32):3000-3008. doi: 10.1200/JCO.18.02306. Epub 2019 Sep 26. PMID 31557067
- [Derived] Leiter U, Stadler R, Mauch C, Hohenberger W, Brockmeyer N, Berking C, Sunderkotter C, Kaatz M, Schulte KW, Lehmann P, Vogt T, Ulrich J, Herbst R, Gehring W, Simon JC, Keim U, Martus P, Garbe C; German Dermatologic Cooperative Oncology Group (DeCOG). Complete lymph node dissection versus no dissection in patients with sentinel lymph node biopsy positive melanoma (DeCOG-SLT): a multicentre, randomised, phase 3 trial. Lancet Oncol. 2016 Jun;17(6):757-767. doi: 10.1016/S1470-2045(16)00141-8. Epub 2016 May 5. PMID 27161539